CLINICAL TRIAL: NCT04034173
Title: FIRE-5 -Study: Optimal Anti-EGFR Treatment of mCRC Patients With Low-Frequency RAS Mutation
Brief Title: Optimal Anti-EGFR Treatment of mCRC Patients With Low-Frequency RAS Mutation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Amgen (Industry); ClinAssess GmbH (Industry)
Responsible Party: Principal Investigator, PD Dr. med. Volker Heinemann, Director of the CCC-Munich at the LMU Munich, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIRE-5
Record Dates: First submitted 2019-01-22; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Treatment Related Cancer
Keywords: colorectal cancer; FIRE; low-RAS; mCRC; Panitumumab
MeSH Terms: conditions — Neoplasms, Second Primary; Colorectal Neoplasms | interventions — Panitumumab; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RAS mutations frequency <= 7% (Other): Panitumumab 6 mg/kg BW as 60-min i.v. infusion* D1
  *If the 1st infusion is well tolerated, all subsequent infusions can be applied over 30-60 minutes.
  Followed by FOLFIRI regimen
  * Irinotecan 180 mg/m² BSA i.v., 30 - 90 min D1
  * Folinic acid (racemic) 400 mg/m²BSA i.v., 120 min D1
  * 5-FU 400 mg/m² BSA, bolus, D1
  * 5-FU 2400 mg/m² BSA i.v. infusion over a period of 46 h D1-2
  q day 14
  Interventions: Drug: Panitumumab; Drug: Irinotecan; Drug: Folinic acid; Drug: 5-FU
- RAS mutation frequency >7% to <=14% (Other): Panitumumab 6 mg/kg BW as 60-min i.v. infusion* D1
  *If the 1st infusion is well tolerated, all subsequent infusions can be applied over 30-60 minutes.
  Followed by FOLFIRI regimen
  * Irinotecan 180 mg/m² BSA i.v., 30 - 90 min D1
  * Folinic acid (racemic) 400 mg/m²BSA i.v., 120 min D1
  * 5-FU 400 mg/m² BSA, bolus, D1
  * 5-FU 2400 mg/m² BSA i.v. infusion over a period of 46 h D1-2
  q day 14
  Interventions: Drug: Panitumumab; Drug: Irinotecan; Drug: Folinic acid; Drug: 5-FU
- RAS mutation frequency >14% to <=20% (Other): Panitumumab 6 mg/kg BW as 60-min i.v. infusion* D1
  *If the 1st infusion is well tolerated, all subsequent infusions can be applied over 30-60 minutes.
  Followed by FOLFIRI regimen
  * Irinotecan 180 mg/m² BSA i.v., 30 - 90 min D1
  * Folinic acid (racemic) 400 mg/m²BSA i.v., 120 min D1
  * 5-FU 400 mg/m² BSA, bolus, D1
  * 5-FU 2400 mg/m² BSA i.v. infusion over a period of 46 h D1-2
  q day 14
  Interventions: Drug: Panitumumab; Drug: Irinotecan; Drug: Folinic acid; Drug: 5-FU

INTERVENTIONS:
Drug: Panitumumab — Panitumumab 6 mg/kg BW as 60-min i.v. infusion* D1
  *If the 1st infusion is well tolerated, all subsequent infusions can be applied over 30-60 minutes.
Drug: Irinotecan — Irinotecan 180 mg/m² BSA i.v., 30 - 90 min D1
Drug: Folinic acid — Folinic acid (racemic) 400 mg/m²BSA i.v., 120 min D1
Drug: 5-FU — 5-FU 400 mg/m² BSA, bolus, D1 5-FU 2400 mg/m² BSA i.v. infusion over a period of 46 h D1-2

SUMMARY:
The present hypothesis is that anti-EGFR agents are active in tumors with low-level RAS mutation when the majority of tumor cells is still sensitive. While response rate may be high and may reflect sensitivity to anti-EGFR agents, PFS is anticipated to be shorter than in RAS wild-type patients due to the faster development of resistance when sensitive cells are eradicated and when the RAS-mutant anti-EGFR resistant clones become predominant.

The characteristics of low-level RAS mutant tumors would be:

* Objective response rate (ORR) high (reflecting the sensitive clone)
* Progression-free survival (PFS) short (reflecting the more rapid outgrowth of RAS mutant clones)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, UICC stage IV metastatic adenocarcinoma of the colon or rectum
* Primarily non-resectable metastases or surgical resection refused by the patient
* RAS mutation determined by the local pathology
* Age ≥18
* ECOG performance status 0-2
* Patients suitable for chemotherapy administration
* Patient's written declaration of consent obtained
* Estimated life expectancy > 3 months
* Presence of at least one measurable reference lesion according to the RECIST 1.1 criteria
* Primary tumor tissue available and patient consents to storage and molecular and genetic profiling of tumor material. Molecular profiling of blood samples is optionally performed.
* Adequate bone marrow function:

  * Leukocytes ≥ 3.0 x 109/L with neutrophils ≥ 1.5 x 109/L
  * Thrombocytes ≥ 100 x 109/L
  * Haemoglobin ≥ 5.6 mmol/L (equivalent to 9 g/dL)
* Adequate hepatic function:

  * Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * ALAT and ASAT ≤ 2.5 x ULN (in the presence of hepatic metastases, ALAT and ASAT ≤ 5 x ULN)
* Adequate renal function:

  ▫ Creatinine clearance (calculated according to Cockcroft and Gault) ≥ 50 mL/min
* No previous chemotherapy for metastatic disease. Patient with need of immediate treatment (high tumor load, symptoms) may have received one application of FOLFIRI prior to study treatment.

Exclusion Criteria:

* Previous chemotherapy for metastatic disease with the exception of one cycle of FOLFIRI (e.g. while waiting for the result of RAS mutation frequency).
* Patients planned to be treated with FOLFOX or another oxaliplatin-based regimen as first-line treatment
* Primarily resectable metastases and the patient agrees to resection
* Grade III or IV heart failure (NYHA classification)
* Medical or psychological impairments associated with restricted ability to give consent or not allowing conduct of the study
* Previous chemotherapy for the colorectal cancer with the exception of adjuvant treatment, completed at least 6 months before entering the study
* Participation in an investigational clinical study or experimental drug treatment within 30 days prior to study inclusion or within a period of 5 half-lives of the substances administered in the investigational clinical study or during an experimental drug treatment prior to inclusion in the study, depending on which period is longest
* Known hypersensitivity or allergic reaction to any of the following substances: 5-fluorouracil, folinic acid, panitumumab, irinotecan, and chemically related substances and/or hypersensitivity to any of the excipients of any of the aforementioned substances including known hypersensitivity reactions to monoclonal antibodies NCI CTCAE Grade ≥ 3.
* Known hypersensitivity to Chinese hamster ovary cell (CHO) - cellular products or other recombinant human or humanised monoclonal antibodies
* History of uncontrolled bronchial asthma
* Patients with interstitial pneumonitis or pulmonary fibrosis
* Patients with known brain metastasis
* History of acute or subacute intestinal occlusion or chronic inflammatory bowel disease or chronic diarrhoea
* Symptomatic peritoneal carcinomatosis
* Severe, non-healing wounds, ulcers or bone fractures
* Patients with acute or chronic infection requiring systemic therapy
* Known history of positive testing for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Active or chronic Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive; serologic tests required in patients who receive study treatment).
* Known DPD deficiency (specific screening not required)
* Known glucuronidation deficiency (Gilbert's syndrome);(specific screening not required
* Treatment with sorivudine or brivudine within 28 days before study enrollment or requirement for concomitant antiviral treatment with sorivudine or brivudine
* History of a second primary malignancy during the past 5 years before inclusion in the study or during participation in the study, with the exception of a basal cell or squamous cell carcinoma of the skin or cervical carcinoma in situ, if these were treated curatively.
* Known previous or ongoing alcohol or drug abuse
* Pregnant or breast-feeding patients
* Any other severe concomitant disease or disorder which, in the investigator's opinion, could influence the patient's ability to participate in the study or influence his/her safety during the study or interfere with interpretation of study results
* Both, absent and restricted legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | up to 60 months
  As primary endpoint ORR according to RECIST 1.1 will be evaluated separately for each arm of patients with defined low-frequency RAS mutation

SECONDARY OUTCOMES:
Progression free survival (PFS) | up to 60 months
  PFS, separately for each arm of patients with defined low-frequency RAS mutation
Overall Survival (OS) | up to 60 months
  OS, separately for each arm of patients with defined low-frequency RAS mutation
Investigation of Early Tumor shrinkage (ETS) as an alternative early-on-treatment predictor of treatment efficacy | up to 48 months
  ETS, separately for each group of patients with defined low-frequency RAS mutation
Investigation of Depth of Response (DpR) to define the nadir of tumour response | up to 48 months
  DpR, separately for each arm of patients with defined low-frequency RAS Mutation.

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Modest, PD Dr., Study Chair — Ludwigs Maximilians University Munich
Locations (1):
- Ludwigs Maximialians University, Munich, Germany

IPD SHARING:
Plan to Share IPD: No